CLINICAL TRIAL: NCT06753630
Title: Does Combined Polydeoxyribonucleotide Improve the Outcome of Extensor Muscle Strengthening Exercise with Extracorporeal Shockwave Therapy for Lateral Epicondylitis of Elbow?: a Randomized Controlled Trial
Brief Title: Polydeoxyribonucleotide for Elbow Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jung-Taek Hwang, Professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-100
Record Dates: First submitted 2024-12-02; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Lateral Epicondylitis; Extracorporeal Shockwave Therapy; Muscle Strengthening
Keywords: Polydeoxyribonucleotide
MeSH Terms: conditions — Tennis Elbow | interventions — Extracorporeal Shockwave Therapy; Sodium Chloride; Polydeoxyribonucleotides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (G1): EMSE + ESWT + Saline Injection (Placebo Comparator): Participants in this group will perform extensor muscle strengthening exercises and receive extracorporeal shockwave therapy. Additionally, they will receive a 3mL saline injection at the first outpatient department visit.
  Interventions: Behavioral: Extensor Muscle Strengthening Exercise; Procedure: Extracorporeal Shockwave Therapy; Drug: Saline injection (Octreotide LAR placebo)
- Group 2 (G2): EMSE + ESWT + PDRN Injection (Experimental): Participants in this group will perform extensor muscle strengthening exercises and receive extracorporeal shockwave therapy. Additionally, they will receive a 3mL injection of polydeoxyribonucleotide (PDRN) at the first outpatient department visit.
  Interventions: Behavioral: Extensor Muscle Strengthening Exercise; Procedure: Extracorporeal Shockwave Therapy; Drug: Polydeoxyribonucleotide Injection

INTERVENTIONS:
Behavioral: Extensor Muscle Strengthening Exercise — A series of exercises aimed at strengthening the extensor muscles of the forearm to alleviate symptoms of lateral epicondylitis.
Procedure: Extracorporeal Shockwave Therapy — A non-invasive procedure that uses shockwaves to promote healing and reduce pain in the affected area.
Drug: Saline injection (Octreotide LAR placebo) — A 3mL injection of saline solution used as a placebo in the study.
  Arms: Group 1 (G1): EMSE + ESWT + Saline Injection
Drug: Polydeoxyribonucleotide Injection — A 3mL injection of polydeoxyribonucleotide (5.625mg/3mL) used to enhance the healing process and improve outcomes in lateral epicondylitis treatment.
  Arms: Group 2 (G2): EMSE + ESWT + PDRN Injection

SUMMARY:
The goal of this clinical trial is to investigate the synergistic effect of polydeoxyribonucleotide (PDRN) on extensor muscle strengthening exercise (EMSE) combined with extracorporeal shockwave therapy (ESWT) for treating lateral epicondylitis (LE) of the elbow in adults aged 18 to 65 years. The main questions it aims to answer are:

Does the addition of PDRN improve pain reduction as measured by the Visual Analog Scale (VAS)? Does the addition of PDRN enhance functional outcomes such as the Mayo Elbow Performance Score (MEPS) and Hand Grip Strength Index (HGSI)?

Researchers will compare two groups to see if PDRN provides additional benefits:

Group 1: EMSE + ESWT + saline injection Group 2: EMSE + ESWT + PDRN injection

Participants will:

Perform extensor muscle strengthening exercises Receive extracorporeal shockwave therapy Receive either a saline injection or a PDRN injection at the first outpatient department visit Attend follow-up visits at 6 and 12 weeks for assessments

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 65 years Diagnosed with chronic lateral epicondylitis (LE) of the elbow Willing to perform extensor muscle strengthening exercises Able to attend follow-up visits at 6 and 12 weeks

Exclusion Criteria:

History of elbow surgery Significant trauma to the elbow Current use of corticosteroids for LE Current use of other treatments for LE Pregnant or breastfeeding women Participation in another clinical trial within the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-11-20 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Pain Reduction | Baseline, 6 weeks, 12 weeks
  Pain Reduction as measured by the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst possible pain), with higher scores indicating worse pain.

SECONDARY OUTCOMES:
Functional Improvement | Baseline, 6 weeks, 12 weeks
  Improvement in elbow function as measured by the Mayo Elbow Performance Score (MEPS). This score ranges from 0 to 100, with higher scores indicating better elbow function. The MEPS assesses pain, range of motion, stability, and daily function.
Grip Strength Improvement | Baseline, 6 weeks, 12 weeks
  Increase in hand grip strength as measured by the Hand Grip Strength Index (HGSI). HGSI is calculated as the ratio of affected side hand grip strength (in Newtons, N) to unaffected side hand grip strength (in Newtons, N). The index does not have predefined minimum or maximum values, as it is a relative measure. Higher values indicate greater improvement in grip strength on the affected side relative to the unaffected side.
Common Extensor Tendon Depth Measured by Ultrasonography | Baseline, 6 weeks, 12 weeks
  Common Extensor Tendon Depth (CETD): Changes in common extensor tendon depth (units: millimeters, mm) as measured by ultrasonography. This measure assesses the structural changes in the tendon.
Color Doppler Activity Measured by Ultrasonography | Baseline, 6 weeks, 12 weeks
  Color Doppler Activity (CDA): Changes in color Doppler activity as measured by ultrasonography. This measure assesses the vascular changes in the tendon.
  Changes in CDA as measured by ultrasonography. CDA was graded on a scale from 0 to 4 within a 0.5-cm longitudinal part of the tendon with maximal Doppler activity. The grading criteria are as follows:
  * Grade 0: No activity
  * Grade 1: Single vessel in the region of interest (ROI)
  * Grade 2: <25% of the ROI
  * Grade 3: 25%-50% of the ROI
  * Grade 4: >50% of the ROI

CONTACTS AND LOCATIONS:
Locations (1):
- Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No